CLINICAL TRIAL: NCT00001780
Title: Stimulation of the Human Central and Peripheral Nervous System With a Magnetic Stimulator
Brief Title: Magnetic Stimulation of the Human Nervous System
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980065; 98-N-0065
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Demyelinating Disease; Healthy; Lysosomal Storage Disease; Motor Neuron Disease; Movement Disorder
Keywords: Myelopathy; Demyelination; Leukodystrophy; Motor Neuron Disease; Movement Disorders; Normal Volunteer
MeSH Terms: conditions — Demyelinating Diseases; Lysosomal Storage Diseases; Motor Neuron Disease; Movement Disorders; Spinal Cord Diseases

SUMMARY:
Transcranial Magnetic Stimulation (TMS) is a non-invasive technique to gather information about brain function. It is very useful when studying the areas of the brain related to motor activity (motor cortex, corticospinal tract, spinal cord and nerve roots). The procedure is conducted by transmitting a magnetic signal into the brain to stimulate an area of the body. Electrodes (small pieces of metal taped to areas of the body) are used in order to measure electrical activity. A magnetic signal is sent from a metal instrument held close to the patient's head, to an area of the brain responsible for motor activity of a certain area of the body. The electrodes pick up and record the electrical activity in the muscles.

This study will employ the use of TMS to diagnose neurological disorders that affect the motor cortex or the corticospinal tract. Normal subjects are sometimes studied to investigate normal activity of the nervous system and to train doctors in clinical neurophysiology and electrodiagnostic medicine at the National Institutes of Health (NIH).

DETAILED DESCRIPTION:
This protocol outlines the use of magnetic stimulation as a diagnostic tool in patients with suspected dysfunction of central motor pathways or nerve roots and as a tool to localize and characterize suspected corticospinal abnormalities in neurologic disorders and systemic disorders with neurological manifestations. The protocol is intended for clinical use.

Transcranial magnetic stimulation has been used for diagnosis of neurologic disorders since 1987. The principles of magnetic stimulation and its use for diagnosis are described in current textbooks of clinical neurophysiology as a routine procedure and should be included in the training program for fellows in clinical neurophysiology and electrodiagnostic medicine at NIH.

The magnetic stimuli are to be given as single or paired pulses at repetition rates less than 1 per second.

ELIGIBILITY:
INCLUSION CRITERIA:

Adult patients with weakness or motor dysfunction.

Children and adolescents with corticospinal tract signs.

Normal volunteers, adults.

Normal volunteers, children aged 4-17.

EXCLUSION CRITERIA:

Pregnant women.

Subjects with implanted devices: pacemakers, medication pumps or defibrillators.

Subjects with metal in the cranium except the mouth.

Subjects with intracardiac lines.

Normal subjects with history of seizures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 1998-02; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Eisen AA, Shtybel W. AAEM minimonograph #35: Clinical experience with transcranial magnetic stimulation. Muscle Nerve. 1990 Nov;13(11):995-1011. doi: 10.1002/mus.880131102. PMID 2233862
- [Background] Wassermann EM, Samii A, Mercuri B, Ikoma K, Oddo D, Grill SE, Hallett M. Responses to paired transcranial magnetic stimuli in resting, active, and recently activated muscles. Exp Brain Res. 1996 Apr;109(1):158-63. doi: 10.1007/BF00228638. PMID 8740220
- [Background] Muller K, Homberg V, Lenard HG. Magnetic stimulation of motor cortex and nerve roots in children. Maturation of cortico-motoneuronal projections. Electroencephalogr Clin Neurophysiol. 1991 Feb;81(1):63-70. doi: 10.1016/0168-5597(91)90105-7. PMID 1705221